CLINICAL TRIAL: NCT07140419
Title: A Prospective, Multicenter, Randomized Controlled Trial on the Impact of Coronary CTA Combined With CT-FFR on Diagnosis and Treatment Decisions and Clinical Outcomes in Emergency Patients With Intermediate Risk Chest Pain
Brief Title: Coronary Computed Tomographic Angiography Combined With CT-FFR in Intermediate-Risk Chest Pain Patients.
Acronym: E-CCTA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Beijing Anzhen Hospital (Other); JiNing NO.1 People Hospital (Unknown); Zhun Ge Er Qi Central Hospital (Unknown)
Responsible Party: Principal Investigator, Chuanbao Li, Clinical Professor, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KYLL-202412(XZ)-014-2
Record Dates: First submitted 2025-08-12; First posted 2025-08-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Chest Pain; Coronary Artery Disease; Emergency Department
Keywords: Intermediate Risk Chest Pain; Emergency Department; CCTA; CT-FFR; Coronary Artery Disease
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Emergencies

STUDY DESIGN:
Intervention Model Description: Patients presenting to the emergency department (ED) with chest pain or other symptoms suggestive of acute coronary syndrome (ACS), who have intermediate risk (defined by a HEART score > 3) and no acute myocardial infarction (MI), will be randomized to one of two strategies after providing written informed consent: an initial approach involving coronary computed tomographic angiography (CCTA) or a standard care pathway without early CCTA.
Who Masked: Outcomes Assessor
Masking Description: Prior to outcome adjudication, all relevant documents will be de-identified to exclude any reference to prior coronary computed tomographic angiography (CCTA) results, ensuring evaluators remain blinded to baseline imaging data that could influence objective assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Patients receive early coronary computed tomographic angiography (CCTA) combined with CT-derived fractional flow reserve (CT-FFR) to guide diagnostic and treatment decisions, in addition to standard care.
  Interventions: Diagnostic Test: Coronary computed tomographic angiography with CT - derived fractional flow reserve
- Control Arm (No Intervention): Patients receive standard care without early CCTA, with further management determined at the discretion of their treating physician.

INTERVENTIONS:
Diagnostic Test: Coronary computed tomographic angiography with CT - derived fractional flow reserve — A non-invasive coronary computed tomography angiography (CCTA) protocol that visualizes coronary anatomy to evaluate the presence, location, and severity of atherosclerotic stenosis, coupled with CT-derived fractional flow reserve (CT-FFR) analysis-a computational fluid dynamics method applied to CCTA datasets-to assess the hemodynamic significance of identified stenoses and identify lesions likely to induce myocardial ischemia.
  Arms: Experimental Arm

SUMMARY:
This study aims to investigate the guiding value of coronary CTA combined with CT-FFR in diagnostic and treatment decision-making for emergency chest pain patients at moderate risk, as well as its impact on clinical outcomes. Through a prospective multicenter randomized controlled trial, this research compares the preventive effects of early application of this technology versus standard care on major adverse cardiovascular events (MACE), with the goal of optimizing the diagnostic and treatment processes for emergency chest pain patients.

DETAILED DESCRIPTION:
This study involves intermediate-risk emergency department patients presenting with chest pain or symptoms suggestive of acute coronary syndrome (ACS) but without acute myocardial infarction (AMI), defined by a HEART score greater than 3. After providing written informed consent, these patients are randomized to one of two strategies: an initial approach incorporating early coronary computed tomographic angiography (CCTA) or a standard care pathway without early CCTA. Patients in the CCTA group receive standard care as determined by their treating physician and undergo CCTA as soon as possible, typically within 24 hours and at most within 21 days. The results of the CCTA, including coronary artery stenosis severity and CT-derived fractional flow reserve (CT-FFR) values, are provided to the physician to inform further management, which may include invasive coronary angiography, medical therapy, or lifestyle interventions.

In contrast, patients randomized to the standard care group without early CCTA proceed with physician-directed evaluations that may include non-invasive functional tests such as exercise electrocardiography, stress echocardiography, or nuclear imaging according to local clinical practices, though CCTA is not part of their initial workup. Both groups receive optimal preventive care in line with current guidelines, and treating physicians are encouraged to initiate secondary prevention measures like antiplatelet therapy or statin use if any diagnostic tests reveal signs of coronary artery disease (CAD).

The primary endpoint of the study is a composite of death, readmission due to myocardial infarction, or hospitalization for unstable angina requiring revascularization. The trial aims to determine whether an early CCTA strategy improves diagnostic and treatment decision-making for intermediate-risk chest pain patients, ultimately influencing clinical outcomes compared to standard care. The study incorporates a prospective, multicenter design to ensure broad applicability and rigor, with careful attention to patient safety and adherence to ethical standards throughout the enrollment and follow-up processes.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years；
2. Within 24 hours of presenting to the emergency department (ED) with chest pain or other symptoms suggestive of coronary artery disease (CAD)；
3. HEART-score >3 (according to http://www.heartscore.nl/)；
4. Signed written informed consent.

Exclusion Criteria:

1. Inability to obtain informed consent；
2. Acute Coronary Syndromes (ACS) requiring urgent revascularization；
3. Known Obstructive Coronary Artery Disease (CAD) or previous PCI or CABG;
4. Concomitant severe congestive heart failure (New York Heart Association [NYHA] class III-IV or left ventricular ejection fraction [LVEF] < 30%) or acute pulmonary edema;
5. Severe hepatic insufficiency (Child-Pugh score ≥ C, or aspartate aminotransferase [AST] > 5× upper limit of normal); severe renal insufficiency (estimated glomerular filtration rate [eGFR] ≤ 30 mL/min/1.73 m²) or patients receiving continuous renal replacement therapy, hemodialysis, or peritoneal dialysis;
6. History of prior coronary artery bypass grafting (CABG);
7. Severe allergy to iodinated contrast agents;
8. Inability to obtain high-quality imaging;
9. Pregnant or lactating females;
10. Concomitant diseases or limited life expectancy, quality of life, or functional status precluding further CAD evaluation;
11. Any other factors that, in the investigator's judgment, make the patient unsuitable for study enrollment, completion of the study, or follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2032-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major adverse cardiovascular events (MACE), defined as the composite endpoint of cardiovascular death, nonfatal myocardial infarction, nonfatal stroke, coronary revascularization, and unstable angina pectoris | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
  Major adverse cardiovascular events (MACE), a pivotal composite endpoint in cardiovascular clinical trials, are defined as the aggregate occurrence of cardiovascular death, nonfatal ST - elevation or non - ST - elevation myocardial infarction (reflecting ischemic myocardial injury), nonfatal ischemic or hemorrhagic stroke (denoting cerebrovascular ischemia or hemorrhage), coronary revascularization (encompassing percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG] for obstructive coronary lesions), and unstable angina pectoris (characterized by new - onset or crescendo chest pain indicative of acute coronary syndrome without myocardial necrosis).

SECONDARY OUTCOMES:
Short-term hospitalization rate | 1 month
Incidence of All-cause mortality | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
  All-cause mortality (cardiovascular death, non-cardiovascular death, death of undetermined cause)
Incidence of Cardiovascular Death | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
Incidence of Nonfatal Myocardial Infarction | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
Incidence of Nonfatal Stroke | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
Incidence of Recurrent Emergency Department Visit for Chest Pain | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled
  Re-presentation with chest pain as the main complaint
Proportion of Patients Undergoing Invasive Coronary Angiography | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
Proportion of Patients with Non-Obstructive CAD at Invasive Coronary Angiography | The enrollment phase will last for 2 years, and follow-up for all participants will continue until 12 months after the last participant is enrolled.
Effect of an Early CCTA with CT-FFR Diagnostic Strategy on Preventive Medication Utilization in Intermediate-Risk Emergency Department Chest Pain Patients | 1 Year, 2 Year, 3 Year, 4 Year, and 5 Year.
  Utilization of preventive medications (based on dispensed prescriptions), including antiplatelet therapy, statins, and antihypertensive agents.
Total Direct Medical Costs per Participant | 1 Year and 5 Year
  Cumulative direct medical costs including emergency department care, diagnostic testing, preventive/therapeutic medications, invasive procedures, and hospitalizations related to cardiovascular events. Costs will be standardized to 2025 Chinese Yuan using national health service price indices.
Quality of Life Assessed by the Seattle Angina Questionnaire (SAQ) | 1 Year and 5 Year
  The Seattle Angina Questionnaire (SAQ) is a validated, patient-reported instrument assessing functional status and quality of life in patients with coronary artery disease. Scores range from 0 to 100, with higher scores indicating better health status and quality of life. Change from baseline to follow-up will be measured.
Quality of Life Assessed by the EQ-5D Index Scores | 1 Year and 5 Year
  The EuroQol 5-Dimension (EQ-5D) questionnaire is a standardized instrument for measuring generic health status. The EQ-5D index score ranges from -0.594 (worst health state) to 1.0 (perfect health). Higher scores indicate better health utility. Change from baseline to follow-up will be measured.

OTHER OUTCOMES:
Number of Participants with Allergic Reactions or Anaphylaxis within 24 Hours Post-CCTA or Invasive Coronary Angiography | Within 24 hours of CCTA or invasive coronary angiography
  Safety Outcome Measure
Number of Participants with Acute Liver or Kidney Injury within 7 Days Post-CCTA or Invasive Coronary Angiography | Within 7 days of CCTA or invasive coronary angiography
  Safety Outcome Measure
Radiation Dose from Coronary Computed Tomography Angiography as Measured by Dose-Length Product (DLP) | Perioperative/Periprocedural
  Safety Outcome Measure

CONTACTS AND LOCATIONS:
Locations (1):
- Chuanbao Li, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gulati M, Levy PD, Mukherjee D, Amsterdam E, Bhatt DL, Birtcher KK, Blankstein R, Boyd J, Bullock-Palmer RP, Conejo T, Diercks DB, Gentile F, Greenwood JP, Hess EP, Hollenberg SM, Jaber WA, Jneid H, Joglar JA, Morrow DA, O'Connor RE, Ross MA, Shaw LJ. 2021 AHA/ACC/ASE/CHEST/SAEM/SCCT/SCMR Guideline for the Evaluation and Diagnosis of Chest Pain: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Nov 30;144(22):e368-e454. doi: 10.1161/CIR.0000000000001029. Epub 2021 Oct 28. PMID 34709879
- [Background] Hoffmann U, Truong QA, Schoenfeld DA, Chou ET, Woodard PK, Nagurney JT, Pope JH, Hauser TH, White CS, Weiner SG, Kalanjian S, Mullins ME, Mikati I, Peacock WF, Zakroysky P, Hayden D, Goehler A, Lee H, Gazelle GS, Wiviott SD, Fleg JL, Udelson JE; ROMICAT-II Investigators. Coronary CT angiography versus standard evaluation in acute chest pain. N Engl J Med. 2012 Jul 26;367(4):299-308. doi: 10.1056/NEJMoa1201161. PMID 22830462
- [Background] Gongora CA, Bavishi C, Uretsky S, Argulian E. Acute chest pain evaluation using coronary computed tomography angiography compared with standard of care: a meta-analysis of randomised clinical trials. Heart. 2018 Feb;104(3):215-221. doi: 10.1136/heartjnl-2017-311647. Epub 2017 Aug 30. PMID 28855273
- [Background] Foy AJ, Dhruva SS, Peterson B, Mandrola JM, Morgan DJ, Redberg RF. Coronary Computed Tomography Angiography vs Functional Stress Testing for Patients With Suspected Coronary Artery Disease: A Systematic Review and Meta-analysis. JAMA Intern Med. 2017 Nov 1;177(11):1623-1631. doi: 10.1001/jamainternmed.2017.4772. PMID 28973101
- [Background] SCOT-HEART Investigators; Newby DE, Adamson PD, Berry C, Boon NA, Dweck MR, Flather M, Forbes J, Hunter A, Lewis S, MacLean S, Mills NL, Norrie J, Roditi G, Shah ASV, Timmis AD, van Beek EJR, Williams MC. Coronary CT Angiography and 5-Year Risk of Myocardial Infarction. N Engl J Med. 2018 Sep 6;379(10):924-933. doi: 10.1056/NEJMoa1805971. Epub 2018 Aug 25. PMID 30145934
- [Background] Moss AJ, Williams MC, Newby DE, Nicol ED. The Updated NICE Guidelines: Cardiac CT as the First-Line Test for Coronary Artery Disease. Curr Cardiovasc Imaging Rep. 2017;10(5):15. doi: 10.1007/s12410-017-9412-6. Epub 2017 Mar 27. PMID 28446943
- [Background] Goodacre S, Thokala P, Carroll C, Stevens JW, Leaviss J, Al Khalaf M, Collinson P, Morris F, Evans P, Wang J. Systematic review, meta-analysis and economic modelling of diagnostic strategies for suspected acute coronary syndrome. Health Technol Assess. 2013;17(1):v-vi, 1-188. doi: 10.3310/hta17010. PMID 23331845
- [Background] Mowatt G, Cummins E, Waugh N, Walker S, Cook J, Jia X, Hillis GS, Fraser C. Systematic review of the clinical effectiveness and cost-effectiveness of 64-slice or higher computed tomography angiography as an alternative to invasive coronary angiography in the investigation of coronary artery disease. Health Technol Assess. 2008 May;12(17):iii-iv, ix-143. doi: 10.3310/hta12170. PMID 18462576
- [Background] Ljung L, Lindahl B, Eggers KM, Frick M, Linder R, Lofmark HB, Martinsson A, Melki D, Sarkar N, Svensson P, Jernberg T. A Rule-Out Strategy Based on High-Sensitivity Troponin and HEART Score Reduces Hospital Admissions. Ann Emerg Med. 2019 May;73(5):491-499. doi: 10.1016/j.annemergmed.2018.11.039. Epub 2019 Jan 17. PMID 30661856
- [Background] Shen C, Ge J. Epidemic of Cardiovascular Disease in China: Current Perspective and Prospects for the Future. Circulation. 2018 Jul 24;138(4):342-344. doi: 10.1161/CIRCULATIONAHA.118.033484. No abstract available. PMID 30571361